CLINICAL TRIAL: NCT02048202
Title: Effects of Medical Clowning (Dream Doctors) on the Development of the Nervous System and the Relationship Between Preterm Premature Baby Parents and NICU Staff
Brief Title: Medical Clowning in the NICU (Neonatal Intensive Care Unit and Their Effects on Parents and Staff
Acronym: clowns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: 38-2013.CTIL
Record Dates: First submitted 2014-01-21; First posted 2014-01-29 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-01

CONDITIONS: Premature Neonate
Keywords: clown; neonate; premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- premature neonate: premature neonate

SUMMARY:
The study will compare intervention by Infant Aquatics to infant massage. The intervention in both methods will start at 36 weeks gestational age for 3 months and will consist of sessions with a therapist every 2 weeks. Development will be assessed and compared at 3, 8 and 18 months using Infant Motor Pattern method, Griffith developmental scales and Vineland adaptive behavior scales.

DETAILED DESCRIPTION:
Preterm infants, a continuously growing population, are at high risk for neurodevelopment impairments ranging from minor neurological dysfunction (MND) to cerebral palsy (CP), mainly due to developmental brain injury. Infant Aquatics have been found to benefit and promote infant development. The support and sensory stimulation of the water may improve the development the sensory, motor, as well as, autonomic system of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* neonates wherein their parents have expressed consent to participate in trail
* neonates with parents who are able to understand and fill in questioners
* neonates with no chromosomal deficiencies and no genetic deficiency

Exclusion Criteria:

* neonates with parents who are unable to understand and fill in questioners
* neonates with intraventricular bleeding IVH/PVH
* neonates with periventricular hemorrhage
* neonates with known chromosomal deficiencies or genetic deficiency

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature neonates 32 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
◦Developmental assessment - a composite of several measures | ◦Time Frame: 3 month

SECONDARY OUTCOMES:
Developmental assessment - a composite of several measures | ◦◦Time Frame: 18 month
  Safety Issue?: No

CONTACTS AND LOCATIONS:
Overall Officials: Shay Barak, MD, Principal Investigator — The Baruch Padeh Medical Center - Poria; Amir Kushnir, MD, Study Chair — The Baruch Padeh Medical Center - Poria; Hagit Friedman, PhD, Principal Investigator — University of Haifa
Locations (1):
- The Baruch Padeh Medical Center - Poria, Tiberias, Israel